CLINICAL TRIAL: NCT01867138
Title: Clinical Outcome of Newborn Infants With Suspected Nosocomial Coagulase-negative Staphylococcal Sepsis Treated With Cefazolin or Vancomycin. A Non-inferiority, Randomized, Controlled Trial
Brief Title: Neonatal Suspected Sepsis Treated With Cefazolin or Vancomycin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Jose Ceriani Cernadas M.D., M.D., Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 563
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Nosocomial Neonatal Sepsis
Keywords: Coagulase negative staphylococcus; nosocomial neonatal sepsis; cefazolin; vancomycin; newborn
MeSH Terms: interventions — Cefazolin; Vancomycin; Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefazolin group (Experimental): Initial empirical treatment with cefazolin and amikacin
  Interventions: Drug: Cefazolin; Drug: Amikacin
- Vancomycin (Active Comparator): Initial empirical treatment with vancomycin and amikacin
  Interventions: Drug: Vancomycin; Drug: Amikacin

INTERVENTIONS:
Drug: Cefazolin
  Arms: Cefazolin group
Drug: Vancomycin
  Arms: Vancomycin
Drug: Amikacin

SUMMARY:
The objective is to evaluate the effectiveness of empiric treatment with cefazolin versus to vancomycin in newborn infants with presumptive clinical signs of hospital acquired bacterial sepsis probably caused by Coagulase-negative staphylococcus.

The investigators hypothesized that newborn infants with the presumptive diagnosis of nosocomial sepsis who received cefazolin as empiric treatment would have a clinical outcome not inferior to that of those treated with vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants older than three days of life with suspected bacterial sepsis and according to attending physicians, with an indication for initial treatment with vancomycin and at least one blood culture taken prior to receiving the antimicrobial treatment.

Exclusion Criteria:

* previous treatment with vancomycin during the week before,
* infants referred from other hospitals and, upon admission, were being treated with antibiotics.

Ages: 4 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Clinical outcome of infants | Seven to ten days after starting antibiotics
  Examination of each newborn infant by two of the investigators independently to establish whether the clinical outcome was adequate or inadequate. In order to achieve greater objectivity, the clinical examination was performed using the following criteria:
  Adequate: when the newborn infant had normal clinical parameters, a good general condition, appropriate tolerance to gastric feeding, normal temperature , negative blood and CSF cultures, and normalized results for the lab tests performed at the onset of the treatment.
  Inadequate: when one or more of the following were present: clinical course with persistence of any of the signs of sepsis, positive blood or CSF cultures after 72 hours from the onset of treatment, persistence of abnormal lab tests, and death by sepsis.

SECONDARY OUTCOMES:
Percentage of infants initially assigned to cefazolin group that were switched to vancomycin. | Within 72 hours of starting treatment
  Patients with an inadequate 72 hour response to cefazolin were crossed over to receive vancomycin. The adjudication of response at 72 hours was delineated in a well-defined algorithm. To minimize bias, the final decision to switch treatments, initiated by the pediatrician in charge, required secondary review and agreement of another participating investigator as well as the attending NICU physician.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Cernadas, M.D., Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Capital, Argentina